CLINICAL TRIAL: NCT07342504
Title: Better Experiences in Substance Treatment: A Brief Alcohol-Focused Intervention Tailored for Patients in Opioid Agonist Treatment
Acronym: Project BEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ND24-05-8578; K23AA029729 (NIH)
Record Dates: First submitted 2026-01-13; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder; Opioid Use Disorder; Alcohol Use; Opioid Use
Keywords: Alcohol Use Disorder; Alcohol Use Disorder (AUD); Cognitive Behavioral Therapy; Opioid Use Disorder; Opioid Use Disorder (OUD); Motivational Enhancement Therapy; Cognitive Behavior Therapy (CBT)
MeSH Terms: conditions — Alcoholism; Opioid-Related Disorders; Alcohol Drinking | interventions — Ethanol; Therapeutics

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive the brief opioid-informed treatment or treatment as usual.
Who Masked: Participant, Outcomes Assessor
Masking Description: PI Carpenter and study therapists will be blinded to assessment outcomes, and assessment RAs will be blinded to participant condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (No Intervention): No intervention is administered. All participants in this study receive prescribed buprenorphine for opioid use disorder and may, related to this, receive behavioral intervention focused on medication adherence and preventing opioid relapse. Treatment As Usual refers to receiving this and no additional intervention.
- Experimental: Brief opioid-informed alcohol treatment (Experimental): The brief opioid-informed alcohol treatment is based upon principles of Motivation Enhancement Therapy (MET) and Cognitive Behavioral Therapy (CBT) tailored to the needs of patients in opioid treatment. Delivered once per week for 4 weeks.
  Interventions: Behavioral: Brief opioid-informed alcohol treatment

INTERVENTIONS:
Behavioral: Brief opioid-informed alcohol treatment — The brief opioid-informed alcohol treatment is based upon principles of Motivation Enhancement Therapy (MET) and Cognitive Behavioral Therapy (CBT) tailored to the needs of patients in opioid treatment. Participants will attend weekly in-person sessions for four weeks.
  Arms: Experimental: Brief opioid-informed alcohol treatment

SUMMARY:
This study will help determine the feasibility and acceptability of a brief opioid-informed alcohol intervention in patients receiving prescribed buprenorphine for opioid use who are currently drinking alcohol. It will also provide initial information on whether the intervention improves outcomes related to alcohol use. The results of this proof-of-concept study will inform whether a future larger clinical trial is warranted.

DETAILED DESCRIPTION:
Alcohol use is an under-recognized contributor to the ongoing opioid overdose epidemic, increasing the risk of overdose when used together with opioids. Further, alcohol use and related problems are prevalent among patients in opioid agonist treatment (OAT) and increase the risk of opioid relapse and early departure from treatment. Office-based buprenorphine treatment, a fast-growing form of OAT, is effective at treating opioid use disorder and decreasing risk of opioid overdose, but relapse rates are high in the first year of treatment. There is a significant need to improve treatment retention. Reducing alcohol use and use-related problems in patients receiving buprenorphine may have a significant indirect effect on improving buprenorphine outcomes. However, minimal existing work has examined alcohol interventions in this population. Of the few studies that have, all of them tested standard alcohol interventions that were not tailored to the unique circumstances of opioid treatment or the needs of individuals in OAT. The purpose of this study is to examine the feasibility and acceptability of a brief opioid-informed alcohol intervention and whether the intervention can improve alcohol outcomes. The intervention is based upon principles of motivational enhancement therapy and cognitive behavioral therapy and tailored to the needs of patients receiving OAT.

ELIGIBILITY:
Inclusion Criteria for the RCT:

* Participants must be taking prescribed buprenorphine for at least 2 weeks
* Participants must be 18 years or older.
* Meet DSM-5 criteria for alcohol use disorder (AUD)
* Participants must report alcohol use ≥ 1 day/week on average in the past 28 days
* Participants must be able to read simple English

Exclusion Criteria:

* Currently receiving formal alcohol use treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-21 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the treatment | Assessed at Week 4 (end of trial)
  Acceptability will be assessed with the Satisfaction Questionnaire (CSQ-8), which ranges in scores from 8 to 32 (higher scores indicate higher satisfaction). Treatment satisfaction will be considered acceptable if the number and percentage of subjects who rate their treatment experience in the "satisfactory" or "highly satisfactory" range on the CSQ-8 is ≥ 80%.
Feasibility of the treatment | Assessed at Week 4 (end of trial)
  Retention feasibility will be determined by the number and percentage of enrolled participants who complete the four week treatment protocol.

OTHER OUTCOMES:
Alcohol Use Quantity | Change from baseline to end of treatment (week4), 1-, and 3-month follow up.
  Assessed using Timeline Followback. Typical weekly drinking quantity estimates will be summed to create a "drinks per week" total score, which will be used as our outcome variable.
Buprenorphine Treatment Status | Change from baseline to end of treatment (week4), 1-, and 3-month follow up.
  Whether the participant reports that they are currently receiving prescribed buprenorphine.
Alcohol-related consequences | Change from baseline to end of treatment (week4), 1-, and 3-month follow up.
  Assessed using the Drinker Inventory of Consequences-Recent (DrINC-2R). Common, moderately common, and rare consequences will be examined separately.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Notre Dame, Notre Dame, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Per sponsor requirements, all data will be uploaded to the NIAAA Data Repository.
Time Frame: One year after the completion of the project.
Access Criteria: As required by the Sponsor, the data from this clinical trial will be uploaded to the National Institute on Alcohol Abuse and Alcoholism (NIAAA) data repository. Like all NIAAA grants, the NIAAA will govern the access criteria.

DOCUMENTS (1):
  • Informed Consent Form (2026-01-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT07342504/ICF_000.pdf